CLINICAL TRIAL: NCT03115034
Title: The Protective Effect of Melatonin in Patients Under Carotid Endarterectomy
Brief Title: Melatonin in Patients Under Carotid Endarterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LCW-ZS1057
Record Dates: First submitted 2017-03-22; First posted 2017-04-14 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-03

CONDITIONS: Carotid Stenosis
Keywords: carotid stenosis; melatonin; vascular injury; ischemia reperfusion
MeSH Terms: conditions — Carotid Stenosis; Vascular System Injuries | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CEA with melatonin (Active Comparator): Patients under CEA with melatonin taken during perioperative period.
  Interventions: Drug: Melatonin
- CEA with placebo (Placebo Comparator): Patients under CEA with placebo taken during perioperative period.
  Interventions: Drug: placebo
- CEA with blank control (Sham Comparator): Patients under CEA with nothing unnecessary taken during perioperative period.
  Interventions: Other: blank

INTERVENTIONS:
Drug: Melatonin — Patients under CEA taking 6mg/day melatonin orally from 3 days before operation to 3 days after operation.
  Arms: CEA with melatonin
Drug: placebo — Patients under CEA taking placebo orally from 3 days before operation to 3 days after operation.
  Arms: CEA with placebo
Other: blank — Patients under CEA without taking melatonin or placebo
  Arms: CEA with blank control

SUMMARY:
The main purpose of this study is to evaluate the effects of melatonin in the regulation of the vascular injury in patients under carotid endarterectomy through population-based, randomized, double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
Trial Title: The protective effect of melatonin in patients under carotid endarterectomy Protocol: Investigators recruited eligible Han Chinese participants (aged 40-80) who were diagnosed with carotid stenosis and had indications for carotid endarterectomy (CEA). Participants were excluded if participants had undergone surgical contraindication, or cardiovascular disease, or cerebral infarction within 3 months, or psychiatric disorders, or cancer, or pregnant, or lactating, or taking antipsychotic drugs during perioperative period. Participants were randomly divided into groups of CEA with oral melatonin, CEA with oral placebo, and CEA with blank control. Participants in groups of CEA with oral melatonin and CEA with oral placebo took melatonin orally 6mg/day or placebo from 3 days before operation to 3 days after operation. Blood samples (about 3 milliliter) were taken at baseline, 6h after the operation and 24h after the operation. Through a series hospital clinical laboratory and related ELISA kits to detect endothelial cell injury and ischemia reperfusion in serum markers. Superoxide dismutase (SOD), malonaldehyde (MDA), S100B protein, endothelial nitric oxide synthase (eNOS), nuclear erythroid 2-related factor 2 (Nrf - 2), Interleukin 6 (IL-6), nuclear transcription factor κB p65 (NF-κB p65) were included for analysis to verify whether melatonin have protective effect in patients under carotid endarterectomy. This trial is approved by the Ethical Committee of Peking Union Medical College Hospital (No ZS 1057). All participants completed a questionnaire and signed an informed consent document. Otherwise, participants will get appropriate economic compensation. To achieve treatment concealment, melatonin and placebo in appearance and package were identically. Trial associates monitored compliance with the masking procedure throughout the trial. All participants and study investigators were unaware of treatment allocation throughout the study. The randomization codes remained sealed until after data collection and cleaning, and completion of a masked analysis. The study team monitored and classified protocol deviations. Investigators summarized baseline clinical and demographic characteristics with descriptive statistics and then determined by the Univariate Analysis of Variance. All the data analyses were done using statistical software SPSS 20.0.

Expected results: Compared with patients under CEA with placebo or blank, patients took melatonin have a lower vascular injury and ischemia reperfusion injury.

Consent document: The potential risk, research as a treatment drug of melatonin may delay the metabolism of antipsychotic antipsychotic drug, so when investigators recruit psychiatric disorders or taking antipsychotic drugs orally during the 2 weeks of the trial should exclusion. As a Health care medicine. Melatonin is not suitable for children, so investigators selected recruiting participants under the age of 40 to 80.

The measure to minimize the risk, fully inform the participants and their families the trial's advantages, disadvantages and desired effect. All participants totally agree with the subjects. In this process, at least three or more effective way to get contact with the medical staff or doctor and ensure that those unexpected accident should deserve effective tackle. Participants guarantee to comply with the criterion before start of the trial. Our research involves the application of melatonin is through the china food and drug administration (CFDA) approved to ensure its safety (include its chemical composition, structure, content parameters, main raw material and appropriate crowd). All staff is qualified medical professionals to guarantee the safety of all participants.

The potential risks or discomfort, or inconvenience, or benefits for participants: So far, effective of melatonin in human include regulating sleep, anti-tumor, immune regulation, regulating of inflammation and immune and regulating blood lipid metabolism is confirmed. Adverse reactions is slow the delay of antipsychotic drug metabolism (so nearly one month ago and during period of the trial participants should not taking antipsychotic drugs) during the trial. The basic principle during the trial is ensure safety of participants.

The relevant content consultation: Everyone have the right to consultation the research content through telephone: +86 01069152500 (principal investigator) and +86 01069155817(Ethics committee).

The rights of withdrew from the trial: Participate in the trial is completely voluntary. If for any reason, participants not willing to participate in, or do not wish to continue to participate in this trial, will not affect the rights and interests of participants. In addition, participants have the right to withdraw this trial at any time. If participants do not according to the doctor instructions, or for the sake of your health and benefits, the doctor or the researchers may also require participants to quit the trial.

The compensation of research: If the participants have any unexpected accident relation with the trial, the compensation and responsibility will be provided by Peking union medical college hospital.

Privacy protection: The privacy of every participant will be protected. The results of the trial in academic publications will not leak any information to identify your personal identity. Peking union medical college hospital will save everybody's data and guarantee not leak without authorization.

Investigators declare no competing interests.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with carotid stenosis
* had indications for carotid endarterectomy (CEA)

Exclusion Criteria:

* surgical contraindication
* cardiovascular disease
* cerebral infarction within 3 months
* psychiatric disorders
* cancer
* pregnant
* lactating
* taking antipsychotic drugs during perioperative period

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Melatonin effects on patients under CEA assessed by the concentration of SOD | 3 months
  Melatonin effects on patients under CEA are detected by the concentration of SOD by ELISA kit.
Melatonin effects on patients under CEA assessed by the concentration of MDA | 3 months
  Melatonin effects on patients under CEA are detected by the concentration of MDA by ELISA kit.
Melatonin effects on patients under CEA assessed by the concentration of S100b | 3 months
  Melatonin effects on patients under CEA are detected by the concentration of S100b by ELISA kit.
Melatonin effects on patients under CEA assessed by the concentration of eNOS | 3 months
  Melatonin effects on patients under CEA are detected by the concentration of eNOS by ELISA kit.
Melatonin effects on patients under CEA assessed by the concentration of Nrf-2 | 3 months
  Melatonin effects on patients under CEA are detected by the concentration of Nrf-2 by ELISA kit.
Melatonin effects on patients under CEA assessed by the concentration of IL-6 | 3 months
  Melatonin effects on patients under CEA are detected by the concentration of IL-6 by ELISA kit.
Melatonin effects on patients under CEA assessed by the concentration of NF-κB p65 | 3 months
  Melatonin effects on patients under CEA are detected by the concentration of NF-κB p65 by ELISA kit.

CONTACTS AND LOCATIONS:
Overall Officials: Changwei Liu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Changwei Liu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kalimeris K, Kouni S, Kostopanagiotou G, Nomikos T, Fragopoulou E, Kakisis J, Vasdekis S, Matsota P, Pandazi A. Cognitive function and oxidative stress after carotid endarterectomy: comparison of propofol to sevoflurane anesthesia. J Cardiothorac Vasc Anesth. 2013 Dec;27(6):1246-52. doi: 10.1053/j.jvca.2012.12.009. Epub 2013 May 30. PMID 23725684
- [Background] Lieb M, Shah U, Hines GL. Cerebral hyperperfusion syndrome after carotid intervention: a review. Cardiol Rev. 2012 Mar-Apr;20(2):84-9. doi: 10.1097/CRD.0b013e318237eef8. PMID 22183061
- [Background] Cheng L, Jin Z, Zhao R, Ren K, Deng C, Yu S. Resveratrol attenuates inflammation and oxidative stress induced by myocardial ischemia-reperfusion injury: role of Nrf2/ARE pathway. Int J Clin Exp Med. 2015 Jul 15;8(7):10420-8. eCollection 2015. PMID 26379832
- [Background] Andersen LP, Rosenberg J, Gogenur I. Perioperative melatonin: not ready for prime time. Br J Anaesth. 2014 Jan;112(1):7-8. doi: 10.1093/bja/aet332. No abstract available. PMID 24318695
- [Background] Wang Z, Ni L, Wang J, Lu C, Ren M, Han W, Liu C. The protective effect of melatonin on smoke-induced vascular injury in rats and humans: a randomized controlled trial. J Pineal Res. 2016 Mar;60(2):217-27. doi: 10.1111/jpi.12305. Epub 2016 Jan 13. PMID 26681403
- [Background] Walsh SR, Nouraei SA, Tang TY, Sadat U, Carpenter RH, Gaunt ME. Remote ischemic preconditioning for cerebral and cardiac protection during carotid endarterectomy: results from a pilot randomized clinical trial. Vasc Endovascular Surg. 2010 Aug;44(6):434-9. doi: 10.1177/1538574410369709. Epub 2010 May 18. PMID 20484064
- [Background] Lapi D, Vagnani S, Cardaci E, Paterni M, Colantuoni A. Rat pial microvascular responses to melatonin during bilateral common carotid artery occlusion and reperfusion. J Pineal Res. 2011 Aug;51(1):136-44. doi: 10.1111/j.1600-079X.2011.00870.x. Epub 2011 Apr 7. PMID 21470301
- [Background] Parsson HN, Lord RS, Scott K, Zemack G. Maintaining carotid flow by shunting during carotid endarterectomy diminishes the inflammatory response mediating ischaemic brain injury. Eur J Vasc Endovasc Surg. 2000 Feb;19(2):124-30. doi: 10.1053/ejvs.1999.0954. PMID 10727360
- [Background] Weigand MA, Laipple A, Plaschke K, Eckstein HH, Martin E, Bardenheuer HJ. Concentration changes of malondialdehyde across the cerebral vascular bed and shedding of L-selectin during carotid endarterectomy. Stroke. 1999 Feb;30(2):306-11. doi: 10.1161/01.str.30.2.306. PMID 9933264
- [Background] Kalra VB, Rao B, Malhotra A. Teaching NeuroImages: perfusion imaging of cerebral hyperperfusion syndrome following revascularization. Neurology. 2013 Jul 23;81(4):e25-6. doi: 10.1212/WNL.0b013e31829c5cae. PMID 23877801
- [Background] Ge YL, Li X, Gao JU, Zhang X, Fang X, Zhou L, Ji W, Lin S. Beneficial effects of intravenous dexmedetomidine on cognitive function and cerebral injury following a carotid endarterectomy. Exp Ther Med. 2016 Mar;11(3):1128-1134. doi: 10.3892/etm.2016.2978. Epub 2016 Jan 11. PMID 26998048
- [Background] Cervantes M, Morali G, Letechipia-Vallejo G. Melatonin and ischemia-reperfusion injury of the brain. J Pineal Res. 2008 Aug;45(1):1-7. doi: 10.1111/j.1600-079X.2007.00551.x. Epub 2008 Jan 9. PMID 18194199